CLINICAL TRIAL: NCT05420805
Title: Protective Effects of Pre- and Post-biotics on Gut Inflammation, Microbiota Diversity, Epileptogenesis, and Quality of Life in Rett Syndrome
Brief Title: Protective Role of Pre-/ Post-biotics on Gut Inflammation, Dysbiosis, and Life Quality in Rett Syndrome (Biotics_RTT)
Acronym: Biotics_RTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Senese (Other)
Collaborators: Kolfarma s.r.l. - Italy (Unknown); European Institute of Oncology (Other)
Responsible Party: Principal Investigator, Claudio De Felice, Principal Investigator, Azienda Ospedaliera Universitaria Senese
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NCT
Record Dates: First submitted 2022-06-13; First posted 2022-06-15 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Rett Syndrome; Dysbiosis; Epilepsy; Quality of Life
Keywords: Gut dysfunction; Inflammation; Alpha-lactalbumin; Butyrate
MeSH Terms: conditions — Rett Syndrome; Dysbiosis; Epilepsy; Inflammation | interventions — Inulin; Butyric Acid; Zinc Oxide

STUDY DESIGN:
Intervention Model Description: This is a 29-week pilot, single site, randomized, cross-over trial of alpha-lactalbumin + sodium butyrate + inulin + fructo-oligosaccharides vs. sodium butyrate + zinc oxide. Periods I and II of the randomized study are 12 weeks long together with a 4 week washout period.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double (Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre- and post-biotic (ALAC, inulin, FOS, and sodium butyrate) (Active Comparator): The product (ALAC+butyrate+inulin+fructo oligosaccharides FOS) is a powder for oral suspension. Dosage is dependent on weight. For participants weighing <50 kg, a 4 g dose (i.e., one 4 g sachet) is intended to be administered orally once a day after dissolving in water. For participants weighing ≥50 kg, a 4 g dose (i.e., 4 g sachets) is intended to be administered orally twice a day (12h interval) after dissolving in water.
  Interventions: Dietary Supplement: ALAC, inulin, FOS, and sodium butyrate
- Post-biotic (sodium butyrate and zinc oxide) (Active Comparator): The product (sodium butyrate+ zinc oxide) is in the form of tablets. Dosage is dependent on weight. For participants weighing <25 kg, one 380 mg tablet is intended to be administered orally twice a day . For participants weighing 25 to 40 kg, three 380 mg tablet dose is intended to be administered orally according to the 2+1 tablets per day schedule (12h interval). For participants weighing ≥40 kg, four 380 mg tablet dose is intended to be administered orally according to the 2+2 tablets per day schedule (12h interval).
  Interventions: Dietary Supplement: Sodium butyrate and zinc oxide

INTERVENTIONS:
Dietary Supplement: ALAC, inulin, FOS, and sodium butyrate — Pre- and post-biotic supplementation will be administered for 3 month period (i.e. 12 weeks) given the filling out of a supplementation diary by parents/caregivers. At the scheduled visits/ phone contacts (i.e., baseline, 4 weeks and 12 weeks), systemic inflammation, intestinal inflammation, and gut microbiome characterization as well as treatment compliance, clinical and dietary intake will be assessed. A seizure diary will be provided to parents/caregivers in order to check the frequency and entity of the critical episodes. An EEG recording will be performed at enrollment (or within 6 months prior to the baseline visit).
  Arms: Pre- and post-biotic (ALAC, inulin, FOS, and sodium butyrate)
Dietary Supplement: Sodium butyrate and zinc oxide — Post-biotic supplementation will be administered for 3 month period (i.e. 12 weeks) given the filling out of a supplementation diary by parents/caregivers. At the scheduled visits/ phone contacts (i.e., baseline, 4 weeks and 12 weeks), systemic inflammation, intestinal inflammation, and gut microbiome characterization, as well as treatment compliance, clinical and dietary intake will be assessed. A seizure diary will be provided to parents/caregivers in order to check the frequency and entity of the critical episodes. An EEG recording will be performed at enrollment (or within 6 months prior to the baseline visit).
  Arms: Post-biotic (sodium butyrate and zinc oxide)

SUMMARY:
The study will examine the potential efficacy and safety of two pre- and post-biotics on markers for gut inflammation and intestinal microbiota ecology in patients with Rett syndrome. Moreover, this trial will search for possible effects on epileptogenesis and quality of life.

DETAILED DESCRIPTION:
The gastrointestinal tract is the major site of exposure to environmental molecules where 1) dietary components are chemically transformed by the microbiota, and 2) gut-derived metabolites are disseminated to all organs, including the brain. The human gut microbiota directly affects human health, and its alteration can lead to gastrointestinal abnormalities and inflammation. Indeed, accumulating clinical and experimental evidences indicate that the gut microbiota impacts behavior, modulates neurotransmitter production in the gut and brain, influences brain development and myelination patterns. Specific gut-derived metabolites, such as 4-ethylphenyl sulfate (4-EPS) and isoamylamine (IAA) are known to alter brains activity and anxiety behavior in mice and/ or promoting neural cell death leading to cognitive decline. Rett syndrome (RTT; Online Mendelian Inheritance in Man, OMIM number #312750) is a severe and progressive neurological disorder that almost exclusively affects females with an incidence of ~1:10,000 live births. Loss-of-function mutations of the X-linked methyl-CpG binding protein 2 (MeCP2) gene is the major cause (approximately 90 %) of classical cases of RTT. Although a rare disorder, RTT represents a leading cause of severe cognitive impairment in the female gender. Affected individuals commonly show a period of apparent early normal development, followed by regression of hand and/or communication skills, and subsequent development of hand stereotypies, while gait is often abnormal in those who are learning to walk.

Despite a wide phenotypic variability, RTT is commonly associated with epilepsy, sleep disturbances, and gastrointestinal dysfunction thus suggesting a link between RTT's gastrointestinal abnormalities and the gut microbiota.

RTT is associated with a dysbiosis of both the bacterial and fungal component of the gut microbiota, suggesting that MeCP2 loss-of-function can favour the establishment of a peculiar microbial community with altered production of short chain fatty acids (SCFAs) possibly contributing to the RTT gastrointestinal physiopathology.

Modulation of the systemic inflammatory response using pre- and post-biotics is advocated as a possible global therapeutic approach in neurological diseases such as Alzheimer's dementia.

Alpha-lactalbumin (ALAC), is the predominant whey protein in human milk, provides essential amino acids for protein synthesis in the developing neonates. Its supplementation in adults are associated with improved cognition, better memory and sleep. The bioactive properties of ALAC relate to antimicrobial activity, pre-biotic features and epithelial restoration via selective apoptosis activity. Moreover, the antibacterial peptides released from ALAC during digestion can exert immunostimulatory effects inducing phagocytic activity. Overall, ALAC shows reduction of inflammation and oxidative stress status as well as improvement of insulin resistance and increase in the synthesis of brain serotonin, a central nervous system neurotransmitter with well-known antiepileptic activity.

Butyrate, a bacterial metabolite and one of the main SCFAs, exhibits a broad range of pharmacological activities including microbiome modulating, anti-inflammatory, metabolic pathway regulating and anti-oxidant actions.

This body of knowledge supports testing pre- and post-biotics strategies for benefit in individuals with Rett syndrome with the goal of translating potential new treatments from experimental models to clinical practice. Results of this study could lead to the first approved pre- / post-biotics treatment for common co-morbidities in the disorder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of classic/typical Rett syndrome (and proven loss-of-function mutation of the MeCP2 gene) with gastrointestinal dysfunction and/or positive history of epilepsy
* Female gender (age > / = 3 years old)
* Ability to obtain written informed consent from their parent(s)/legal guardian(s)
* Stable medications for at least 4 weeks prior to the baseline visit.

Exclusion Criteria:

* Diagnosis not fitting into the Rett syndrome consensus guidelines
* Nonpathogenic MECP2 mutation or mutations in non-MECP2 genes (i.e., cyclin-dependent kinase 5, CDKL5; forkhead box protein G1, FOXG1)
* Male gender
* Percutaneous endoscopic gastrostomy (PEG) tube
* Proven hypersensitivity to one or more components of the dietary supplements (X-biotics)
* Unstable concomitant medications less than 4 weeks prior to enrollment visit.
* Concomitant antibiotic therapy at the enrollment. In the case of antibiotic therapy, a 4-weeks washout period will be undertaken.
* Rejection of the informed consent form by the parents/caregivers and/or lack of compliance to the Study procedures.

Min Age: 3 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 28 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Systemic inflammation | Change at 3 months from baseline of each interventional arm
  Change in circulating pro-inflammatory or change in anti-inflammatory cytokine levels
Gut inflammation | Change at 3 months from baseline of each interventional arm
  Change in fecal calprotectin levels
Gut dysbiosis | Change at 3 months from baseline of each interventional arm
  Change in intestinal microbiota biodiversity

SECONDARY OUTCOMES:
Epileptogenesis | Change at 3 months from baseline of each interventional arm
  Change in frequency and/or severity of epileptic seizures (a seizure diary provided to parents/caregivers at the baseline visit)

OTHER OUTCOMES:
Quality of life and gastrointestinal health | Change at 3 months from baseline of each interventional arm
  Change in well-being indices [Quality of Life Inventory-Disability Questionnaire (QI-Disability), Gastrointestinal Health Questionnaire (GHQ), Bristol Stool Chart (BSC), Rome III scoring, Sleep Disturbance Scale for Children Questionnaire (SDSC)]
  [QI-Disability: lower scores indicate a worse outcome, BSC: type 1-2 indicate constipation, type 3-4 normal, and type 5-7 diarrhea), Rome III scoring: higher scores indicate a worse outcome, SDSC: higher scores indicate a worse outcome]
Quality of life and illness severity | Change at 3 months from baseline of each interventional arm
  Change in clinical severity [Rett Syndrome Behaviour Questionnaire (RSBQ) and Motor Behavioural Assessment Scale (MBAS)] (higher scores of RSBQ and MBAS indicate a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio De Felice, MD, Principal Investigator — Policlinico "S. Maria alle Scotte" Azienda Ospedaliera Universitaria Senese , 53100 Siena, Italy
Locations (1):
- Policlinico "S. Maria alle Scotte" Azienda Ospedaliera Universitaria Senese, Siena, Italy

IPD SHARING:
Plan to Share IPD: No